CLINICAL TRIAL: NCT01422083
Title: Correlation Between Loss of Internal Rotation Range of Motion and Size of the Subacromial Space and the Influence of a Home Stretching Program.
Brief Title: Glenohumeral Internal Rotation Deficit (GIRD)
Acronym: GIRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010/372
Record Dates: First submitted 2011-08-22; First posted 2011-08-23 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Glenohumeral Internal Rotation Deficit (GIRD)

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): This group of athletes do not perform a 6-week stretching program.
- Home stretching program (Experimental): These athletes take on a home stretching program (sleeper's stretch).
  Interventions: Procedure: home stretching program

INTERVENTIONS:
Procedure: home stretching program — A home stretching program (sleeper's stretch): 3 x 30 seconds, once a day for 6 weeks.
  Arms: Home stretching program

SUMMARY:
A loss of mobility in the shoulder in direction of internal rotation is associated with shoulder tendon pathology. Cause-effect relationship between these two is still not clear. It is suspected that this loss of mobility reduces the size of the tunnel in which this shoulder tendon is lying, namely the subacromial space. Overhead athletes frequently show glenohumeral internal rotation deficit (GIRD) while being healthy and free of shoulder pain. This makes this population interesting to investigate. This study wants to look at shoulders of overhead athletes with GIRD and measure the size of the subacromial space. After this, the athletes will be instructed to perform a home stretching program and at the end the effect of this on mobility and the size of the subacromial space will be measured.60 athletes will be recruited and randomly allocated to the control group and the stretching group. Before they start stretching, subacromial space size will be measured by use of ultrasound. This is a safe and non-invasive measuring tool. Mobility will be measured by use of a digital inclinometer. This also is safe and non-invasive. Patients will be instructed a stretching exercise, which they will be performing at home once a day during 6 weeks. At the end all outcome measures will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* overhead athletes: at least 3 hours/week training
* male and female
* 18-30 years of age
* No shoulder pain during last 3 months for which a doctor was consulted
* No shoulder surgery
* No neck diseases

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Size of the subacromial space and shoulder mobility. | at 0 weeks
  Measurment of the size of the subacromial space and shoulder mobility are performed by an ultrasound and an inclinometer.
Size of the subacromial space and shoulder mobility. | after 6 weeks
  Measurment of the size of the subacromial space and shoulder mobility are performed by an ultrasound and an inclinometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Cools, Ph.D., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium